CLINICAL TRIAL: NCT05998733
Title: Characteristics of Coagulation in Patients With Sepsis and the Role of Coagulation Disorders in the Development of Disease: a Retrospective Single-center Clinical Study
Brief Title: The Impact of Coagulation Disorders on the Diagnosis and Prognosis of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202300123
Record Dates: First submitted 2023-07-24; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-06

CONDITIONS: Sepsis; Coagulation Disorder
Keywords: sepsis; coagulation disorders
MeSH Terms: conditions — Sepsis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis group: diagnostic sepsis；age>18；Time from clinical symptoms to admission ≤ 7 days； It also meets the following two criteria: ① clinical infection② Sequential Organ Failure Assessment (SOFA) score ≥ 2 points at admission
  Interventions: Diagnostic Test: Early general coagulation function (5 items of coagulation) and thromboelastogram monitoring
- non-sepsis group: diagnostic sepsis；age>18；Time from clinical symptoms to admission ≤ 7 days； It also meets the following two criteria: ① clinical infection②Systemic inflammatory response syndrome(SIRS)，SIRS was defined as the presence of 2 or more of the following: (1) temperature <36℃or >38℃, (2) heart rate >90 beats per minute, (3) respiratory rate >20 breaths per minute or PaCO2 < 32 mm Hg, or (4) white blood cell count ≥12 000 cells/mm3 or≤4000 cells/mm
  Interventions: Diagnostic Test: Early general coagulation function (5 items of coagulation) and thromboelastogram monitoring

INTERVENTIONS:
Diagnostic Test: Early general coagulation function (5 items of coagulation) and thromboelastogram monitoring — * Correlation analysis of sepsis severity with FDP and D-Dimer
  * Discussion on the critical value and area under the curve of FDP and D-Dimer in diagnosis of sepsis
  * Differences in age and sex of FDP and D-Dimer in diagnosis of sepsis
  * Effect of FDP and D-Dimer diagnosis of sepsis on severe conversion rate and all-cause mortality of patients
  * The difference of thromboelastogram in patients with sepsis of different severity
  * Thromboelastogram items (R time α Correlation between angle, k time, maximum blood clot strength and comprehensive coagulation index) and sepsis

SUMMARY:
The study was a retrospective, single-center clinical study. From all patients admitted to the emergency ICU during the period of 2013.1.1-2019.12.31, the investigators screened all patients who met the criteria of 1) ≤7 days from symptom onset to enrollment; 2) patients who also met the criteria of the presence of clinical infections and Sequential Organ Failure Assessment (SOFA) score ≥2; and 3) met the exclusion criteria, and retrospectively collected coagulation indices of the patients before anticoagulation with or without the use of heparin or low molecular heparin, and recorded the worst values of coagulation function of patients before heparin were recorded, and the organ function, inflammatory response, immune indexes, and conversion rate of severe disease were observed, so as to investigate the role of conventional coagulation indexes (FDP, D-dimer) and thromboelastography in the early diagnosis of septicemia patients and to indicate the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Time from clinical symptoms to admission ≤ 7 days；
* infection was diagnosed by clinician
* Systemic inflammatory response syndrome，Systemic inflammatory response syndrome was defined as the presence of 2 or more of the following: (1) temperature <36℃or >38℃, (2) heart rate >90 beats per minute, (3) respiratory rate >20 breaths per minute or PaCO2 < 32 mm Hg, or (4) white blood cell count ≥12 000 cells/mm3 or≤4000 cells/mm

Exclusion Criteria:

* Pregnancy and lactation
* Have hematological diseases (including acute and chronic leukemia, hemolytic anemia, hemophilia, aplastic anemia, bone marrow fibrosis, congenital or acquired coagulation factor deficiency, etc.)
* Anticoagulant or antiplatelet drug treatment
* 24 hours after severe trauma or surgery
* Autoimmune diseases
* cirrhosis
* Malignant tumor patients with personal history or undergoing radiotherapy, chemotherapy and targeted treatment

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study was a retrospective, single-center clinical study. From all patients admitted to the emergency ICU during the period 2013.1.1-2019.12.31, all patients who met the enrollment criteria were screened, and the coagulation function indexes of patients with or without heparin or low molecular heparin before anticoagulation were retrospectively collected, the worst value of coagulation function of patients before heparin was recorded, and the organ function, inflammatory response, immune indexes, and the rate of conversion to severe disease of the patients were observed, so as to To investigate the role of conventional coagulation indices (FDP, D-dimer) and thromboelastography in the early diagnosis and prognosis of patients with sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The plasma concentration of fibrin degradation products(FDP) in ug/ml | within 3 days of admission before the use of anticoagulant drugs
  The plasma concentration of fibrin degradation products(FDP) was assessed after the participant was enrolled within 3 days of admission before the use of anticoagulant drugs
The plasma concentration of DDimer in ug/ml | within 3 days of admission before the use of anticoagulant drugs
  The plasma concentration of DDimer was assessed after the participant was enrolled within 3 days of admission before the use of anticoagulant drugs

CONTACTS AND LOCATIONS:
Overall Officials: Enqiang Mao, PhD, Study Chair — Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- Department of Emergency, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No